CLINICAL TRIAL: NCT04421690
Title: Computerized Cognitive Training in Middle-Aged Adults With Generalized Anxiety Disorder: A Pilot Study (COGMA)
Brief Title: Computerized Cognitive Training in Middle-Aged Adults With Generalized Anxiety Disorder: A Pilot Study
Acronym: COGMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Ashley Curtis, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021943
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: Anxiety; Middle-Aged; Sleep; Cognition; Older Adults
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to cognitive training or trivia training and will complete measures of anxiety, sleep, cognition (objective, self-efficacy), and self-reported arousal at baseline, and post-intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): 8 week computerized cognitive training
  Interventions: Behavioral: Cognitive Training
- Trivia Training (Active Comparator): 8 week computerized trivia training
  Interventions: Behavioral: Trivia Training

INTERVENTIONS:
Behavioral: Cognitive Training — Participants (n=15) will complete computerized cognitive training games and activities online 3 times/week for 8 weeks.
  Arms: Cognitive Training
Behavioral: Trivia Training — Participants (n=15) will receive computerized trivia questions to answer and submit 3 times/week for 8 weeks.
  Arms: Trivia Training

SUMMARY:
The purpose of this research is to look at the effects of computerized cognitive training on anxiety, sleep, mental abilities (cognition), and other aspects of daytime functioning, such as arousal.

ELIGIBILITY:
Inclusion Criteria:

* 45-59 yrs of age
* no neurological or psychiatric illness, dementia, or loss of consciousness > 5 mins
* nongamers (i.e., report <1 hour of video/cognitive training games/week over last 2 yrs)
* proficient in English (reading and writing)
* computer meets technology requirements (i.e. Windows: Windows 7 or above using Internet Explorer 11 or Edge, Mozilla Firefox 41 and above, Google Chrome 48 and above; Mac OS: Mac OS X v10.8 and above using Safari 10 and above, Mozilla Firefox 42 and above, Google Chrome 48 and above; Android App: Android 6 or higher version; iOS App: iOS 10 or higher version
* meet clinical dx criteria for Generalized Anxiety Disorder.

Exclusion Criteria:

* unable to provide informed consent
* unable to undergo randomization
* Telephone Interview for Cognitive Status-modified (TICS) score <33, 2)
* other sleep disorder (i.e., sleep apnea, Periodic Limb Movement Disorder-PLMD, narcolepsy, REM Sleep Behavior Disorder)
* severe untreated psychiatric comorbidity that renders randomization unethical
* psychotropic, anxiolytic medications or other medications(e.g., beta-blockers) that alter mood or sleep
* uncorrected visual/auditory impairments
* participation in nonpharmacological treatment for sleep/fatigue/mood outside the current study.

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Objective Cognition - Computerized Cognitive Tasks | Up to 10 weeks
  Complete computerized tasks. These tasks will measure cognitive functions (e.g., processing speed).
Objective Cognition - Computerized Cognitive Tasks | Up to 10 weeks
  Complete computerized tasks. These tasks will measure cognitive functions (e.g., attention).
Objective Cognition - Computerized Cognitive Tasks | Up to 10 weeks
  Complete computerized tasks. These tasks will measure cognitive functions (e.g., executive function).
Subjective Cognitive Self-Efficacy. -Cognitive Failures Questionnaire | Up to 10 weeks
  A 25-item questionnaire. Participants rate from 0 (never) to 4 (very often) frequency of cognitive errors. Higher scores indicate lower cognitive self-efficacy.
Coronavirus Anxiety Scale | Up to 10 weeks
  5- item questionnaire that assess anxiety related to the Coronavirus.
Anxiety - State-Trait Anxiety Inventory | Up to 10 weeks
  Inventory that asks respondents to rate how true 20 self-descriptive statements (e.g., I feel calm) are on a 4-point scale (1 = not at all, 4 = very much so). Typically, respondents are asked to rate statements according to how they generally feel (trait-anxiety scale) and how they feel in the current moment (state-anxiety scale). Total scores range from 20 to 80, with higher scores indicating greater maladjustment.

SECONDARY OUTCOMES:
Game-related experience- Sessions and duration played | Up to 10 weeks
  During the intervention phase the cognitive training group will play games and will need to log the days and duration played.
Circadian Rhythm- Morningness-Eveningness Questionnaire | Up to 10 weeks
  19-item questionnaire that assesses preference for morning, afternoon, and evening activities. Total score reflects degree of "morningness" or "eveningness" type.
Subjective Arousal- Global Cognitive Arousal-Perceived Stress Scale | Up to 10 weeks
  Perceived Stress Scale is a self-report measure of how life situations are perceived as stressful. The scale consists of 15 items corresponding to everyday situation and participants are asked to rate on a likert scale from 0 (never) to 4 (very often) how often they felt or thought a specific way. Higher scores correspond to higher perceived stress.
Subjective Arousal- Pre-sleep Arousal Scale | Up to 10 weeks
  Pre-sleep Arousal Scale is a 16-item self-report questionnaire comprising both cognitive and somatic manifestations of arousal.
Subjective Arousal- Arousal Predisposition Scale Subjective Arousal- Arousal Predisposition Scale Subjective Arousal- Arousal Predisposition Scale | Up to 10 weeks
  Arousal Predisposition Scale is a 12-item inventory that has been designed to measure the degree to which an individual experiences arousal. Higher scores indicate greater predisposition to arousal.
Game Engagement Questionnaire | Up to 10 weeks
  Questionnaire assessing the experience of the game.
Mood-Depression-Beck Depression Inventory-II | Up to 10 weeks
  21-item inventory that asks respondents to rate on a scale of 0 (no depressive feelings) to 3 (most depressive feelings) their feelings towards various aspects of daily living/situations. Higher total scores indicate worse depressive symptoms.
Alcohol Use - Alcohol Use Disorder Test | Baseline
  10-item questionnaire that assess the frequency of alcohol use and problems associated with alcohol use over the past year.
Physical Activity - International Physical Activity Questionnaire | Up to 10 weeks
  7- item questionnaire assessing the different kinds of physical activities that the participant does as pat of their everyday life.
Personality - Big Five Inventory | Baseline
  10 question assessment measuring personality.
COVID-19 related media exposure and risk questions | Up to 10 weeks
  20- item questionnaire assessing the effects of news and social media on perception of COVID-19.
Subjective Intervention Efficacy- Internet Intervention Utility Questionnaire | Up to 10 weeks
  16- item questionnaire about the use of the intervention.
Computer Proficiency- Computer Proficiency Questionnaire | Baseline
  This questionnaire asks about participants' ability to perform a number of tasks with a computer. Will be examined as a covariate.
Subjective Behavioral Sleep- Insomnia Severity Index | Up to 10 weeks
  Brief self-report measure of current perception of insomnia symptom severity, distress and daytime impairment. Commonly used in insomnia treatment outcome research.
Beck Depression Inventory-2nd Edition | Up to 10 weeks
  21-item inventory that asks respondents to rate on a scale of 0 (no depressive feelings) to 3 (most depressive feelings) their feelings towards various aspects of daily living/situations. Higher total scores indicate worse depressive symptoms.
Subjective Behavioral Sleep - Electronic Daily Sleep Diaries | Up to 10 weeks
  Online diaries completed each morning (~5 mins); diaries measure sleep onset latency, wake time after sleep onset, total sleep time, and sleep quality.
Subjective Behavioral Sleep - Electronic Daily Sleep Diaries | Up to 10 weeks
  Online diaries completed each morning (~5 mins); diaries measure sleep onset latency
Subjective Behavioral Sleep - Electronic Daily Sleep Diaries | Up to 10 weeks
  Online diaries completed each morning (~5 mins); diaries measure wake time after sleep onset
Subjective Behavioral Sleep - Electronic Daily Sleep Diaries | Up to 10 weeks
  Online diaries completed each morning (~5 mins); diaries measure total sleep time
Subjective Behavioral Sleep - Electronic Daily Sleep Diaries | Up to 10 weeks
  Online diaries completed each morning (~5 mins); diaries measure sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Curtis, PhD, Principal Investigator — University of Missouri- School of Medicine
Locations (1):
- University of Missouri, Columbia, Missouri, United States